CLINICAL TRIAL: NCT06510062
Title: Comparative Evaluation of Sustained Acoustic Medicine Device on Circulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-01-2024
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-08

CONDITIONS: Measurement of Circulation on Anatomical Locations of the Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- SAM Ultrasound Device and Diclofenac Patch 1 (Experimental): Patients receive treatment from the SAM Ultrasonic Diathermy Device 1 hour with 2.5% diclofenac ultrasound gel patch on right forearm. The SAM device emits continuous ultrasound at 3-megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Interventions: Device: Sustained Acoustic Medicine; Drug: 2.5% Diclofenac Patches
- SAM Ultrasound Device and Diclofenac Patch 2 (Experimental): Patients receive treatment from the SAM Ultrasonic Diathermy Device 1 hour with 2.5% diclofenac ultrasound gel patch on left forearm. The SAM device emits continuous ultrasound at 3-megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Interventions: Device: Sustained Acoustic Medicine; Drug: 2.5% Diclofenac Patches
- SAM Ultrasound Device and SAM Patch 1 (Experimental): Patients receive treatment from the SAM Ultrasonic Diathermy Device 1 hour with standard ultrasound gel patch on right forearm. The SAM device emits continuous ultrasound at 3-megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Interventions: Device: Sustained Acoustic Medicine
- SAM Ultrasound Device and SAM Patch 2 (Experimental): Patients receive treatment from the SAM Ultrasonic Diathermy Device 1 hour with standard ultrasound gel patch on left forearm. The SAM device emits continuous ultrasound at 3-megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Interventions: Device: Sustained Acoustic Medicine

INTERVENTIONS:
Device: Sustained Acoustic Medicine — The SAM device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity delivering 18,720 Joules of ultrasound per 4 hour treatment.
  Other Names: SAM; Wearable Ultrasound Device; Long Duration Ultrasound; LITUS Device Wearable; Long Duration Low-Intensity Device
  Arms: SAM Ultrasound Device and Diclofenac Patch 1
Device: Sustained Acoustic Medicine — The SAM device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity delivering 18,720 Joules of ultrasound per 4 hour treatment.
  Other Names: SAM; Wearable Ultrasound Device; Long Duration Ultrasound; LITUS Device Wearable; Long Duration Low-Intensity Device
  Arms: SAM Ultrasound Device and Diclofenac Patch 2
Device: Sustained Acoustic Medicine — The SAM device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity delivering 18,720 Joules of ultrasound per 4 hour treatment.
  Other Names: SAM; Wearable Ultrasound Device; Long Duration Ultrasound; LITUS Device Wearable; Long Duration Low-Intensity Device
  Arms: SAM Ultrasound Device and SAM Patch 1
Device: Sustained Acoustic Medicine — The SAM device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity delivering 18,720 Joules of ultrasound per 4 hour treatment.
  Other Names: SAM; Wearable Ultrasound Device; Long Duration Ultrasound; LITUS Device Wearable; Long Duration Low-Intensity Device
  Arms: SAM Ultrasound Device and SAM Patch 2
Drug: 2.5% Diclofenac Patches — Topical pain relief gel worn via SAM patch.
  Arms: SAM Ultrasound Device and Diclofenac Patch 1; SAM Ultrasound Device and Diclofenac Patch 2

SUMMARY:
Comparative Evaluation of Sustained Acoustic Medicine Device on Circulation

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer

Exclusion Criteria:

* Is pregnant/nursing
* Has an active infection, open sores, or wounds in the treatment area
* Has any preexisting extremity circulation condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Blood Flow (Perfusion Unit) | 0 - 1 hour
  Blood Flow Flux through Upper Extremity (Perfusion Unit)
Ultrasound Diathermy (Degrees Centigrade) | 0 - 1 hour
  Temperature Measurement on Body (Degrees Centrigrade)

CONTACTS AND LOCATIONS:
Overall Officials: George K Lewis, PhD, Principal Investigator — ZetrOZ Systems LLC
Locations (1):
- ZetrOZ Systems LLC, Trumbull, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scanzuso A, Hendren T, Egmont M, Zarkar J, Roberge M. Sustained acoustic medicine increases local circulation with a diclofenac delivery patch: a randomized placebo controlled study. Front Med Technol. 2025 Jul 4;7:1552294. doi: 10.3389/fmedt.2025.1552294. eCollection 2025. PMID 40687068